CLINICAL TRIAL: NCT01375088
Title: Phase I Assessing the Preventing and Therapeutic Effect of Propolis in Radiotherapy Induced Mucositis of Head and Neck Cancers
Brief Title: Assessing the Preventing and Therapeutic Effect of Propolis in Radiotherapy Induced Mucositis of Head and Neck Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, ATESSA PAKFETRAT, Associate professor, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 339888
Record Dates: First submitted 2011-06-01; First posted 2011-06-17 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Radiation-induced Mucositis of Oral Mucous Membranes
Keywords: propolis; mucositis; radiotherapy; cancer
MeSH Terms: conditions — Mucositis; Neoplasms | interventions — Propolis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo mouth wash (Placebo Comparator): 10 patients swish & swallow 15 ml placebo mouth wash for at least 5 min from the first session of radiotherapy until the last session
  Interventions: Drug: propolis
- propolis (Active Comparator): 10 patients swish & swallow 15 ml propolis mouth wash for at least 5 min from the first session of radiotherapy until the last session
  Interventions: Drug: propolis

INTERVENTIONS:
Drug: propolis — 15 ml mouth wash 3 times a day for the whole period of radiotherapy for 5 min swish and then swallow

SUMMARY:
The purpose of this study is to determine whether propolis is effective in the treatment and prevention of radiotherapy induced oral mucositis.

DETAILED DESCRIPTION:
Patients with head and neck malignancy with inclusion criteria randomly divide in 2 groups and take the intervention.

ELIGIBILITY:
Inclusion Criteria: - age >15

* need of radiotherapy
* at least half of the mouth in the field of radiation
* dose 50 -70 Gy
* head & neck malignancy

Exclusion Criteria:

* systemic disease
* FBS > 150 WBC > 3000
* history of radiotherapy
* need of chemotherapy
* systemic disease

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
NCI.CTC Scale | 9 month
  we use NCI-CTC scale for patients in 2 groups to assess effect of propolis mouth wash on prevention and treatment of mucositis in patients under radiotherapy.We measured signs(size and sypmtoms) of mucositis by NCI-CTC scale and also we assessed the onset of the mucositis to describe the prevention efficacy of propolis.

SECONDARY OUTCOMES:
hyposalivation scale | 9 month
  we use a scale for patients in 2 groups to assess effect of propolis maouth wash on subjective xerostomy and signs of candidiasis in patiants under radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: arghavan tonkaboni, resident, Principal Investigator — oral medicine dep, dental school, mashhad university of medical science
Locations (1):
- Mashhad University of Medical Science, Mashhad, Khorasan Razavi, Iran